CLINICAL TRIAL: NCT05366829
Title: Tislelizumab Consolidation After Liver-Directed Therapy for Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: BioGene Pharmaceutical Ltd. (Industry); Natera, Inc. (Industry)
Responsible Party: Principal Investigator, Salma Jabbour, MD, Associate Professor, Department of Radiation Oncology, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 072105; Pro2021001725 (Other: Rutgers, The State University of New Jersey)
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Hepatocellular; Liver Cell Carcinoma
Keywords: Liver-Directed Therapy; Tislelizumab; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — tislelizumab

STUDY DESIGN:
Intervention Model Description: This study is a single-arm open-label phase II clinical trial to evaluate safety of the sequence of definitive therapy followed by Tislelizumab in participants with locally advanced unresectable hepatocellular carcinoma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tislelizumab in conjunction with radiation therapy (Experimental): Participants will receive local therapy including TACE+ RT or Ablation (tumors with incomplete ablation) + RT or RT alone (for patients not eligible for TACE or Ablation) and will be screened for eligibility prior to enrollment.
  Once eligibility has been confirmed, Tislelizumab will be started before radiation therapy and will continue after radiation therapy.
  Participants who do not receive Tislelizumab for a total of two cycles will be replaced and interpreted for only toxicity analysis.
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab (also known as BGB A317) is a humanized, immunoglobulin G4 (IgG4)-variant monoclonal antibody against programmed cell death protein-1 (PD-1) under clinical development for the treatment of several human malignancies. Tislelizumab consolidation therapy after radiation therapy can capitalize on the immunomodulatory effect of radiotherapy and improve tumor responses and patient outcomes.

SUMMARY:
The investigators hypothesize that the addition of Tislelizumab after definitive local therapy for locally advanced inoperable Hepatocellular carcinoma (HCC) will synergize with local therapy as well as treat micro metastatic disease and improve one year progression-free survival rates for participants and optimize local control.

DETAILED DESCRIPTION:
Primary Objective:

To determine if consolidation therapy with Tislelizumab following local therapy improves one year progression-free survival in patients with locally advanced, unresectable Hepatocellular carcinoma ( HCC). Progression-free survival (PFS) is defined as the time from first administration of Tislelizumab until the criteria for disease progression is met by response evaluation criteria in solid tumors (RECIST)1.1 or death as a result of any cause, whichever occurs first.

Secondary Objectives:

1. To determine if consolidation therapy with Tislelizumab after definitive therapy improves time to metastatic disease and overall survival (OS) in subjects with localized, inoperable Hepatocellular carcinoma (HCC).
2. To assess objective response rate, disease control rate, duration of response with consolidation therapy with Tislelizumab after local therapy in subjects with localized, inoperable Hepatocellular carcinoma (HCC).
3. To assess the safety profile of Tislelizumab after definitive therapy.
4. To assess biomarker response as measured by Alpha fetoprotein (AFP), should the patient's tumor produce AFP.

Exploratory objectives:

1. To determine the association of the tumor molecular profile from next-generation sequencing (NGS), of the tissue prior to the initiation of therapy with the treatment response.
2. To analyze Circulating tumor DNA (ct DNA) as a biomarker of response to therapy and early detection of disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Each patient eligible to participate in this study must meet all the following criteria:

  1. Written informed consent
  2. Primary diagnosis of HCC, planned to receive radiation, treatment naïve to systemic therapy for HCC, prior TACE permitted
  3. Hepatocellular carcinoma diagnosis by histologic findings and/or imaging criteria of LI-RADS 5
  4. Eastern Cooperative Oncology Group performance status score of 0-2
  5. Age>/=18 years
  6. Child-Pugh class A liver function or B7, BCLC A-C or deemed not a candidate for surgery or liver transplantation
  7. No extrahepatic metastasis detected on CT chest with or without IV contrast, abdomen and pelvis with IV and oral contrast (triphasic-if feasible based on kidney function), or MRI abdomen/liver and chest CT.
  8. Females of childbearing potential must be willing to use a highly effective method of birth control for the duration of the study, and ≥ 6 months after the last dose of tislelizumab, and have a negative urine or serum pregnancy test ≤ 7 days of first dose of study drug
  9. Non-sterile males must be willing to use a highly effective method of birth control for the duration of the study and for ≥ 6 months after the last dose of tislelizumab. Males must agree not to donate or bank sperm during treatment with tislelizumab and for > 6 months after treatment stop.
  10. Must have 1 target lesion measurable in 1 dimension according to RECIST 1.1.
  11. Demonstrate adequate bone marrow and organ function as defined below:

      1. Hematologic - Absolute neutrophil count (ANC) ≥ 1,500/mcL, Hemoglobin > 8.5 g/dL, Platelet count ≥ 75,000/mcL
      2. Renal - Serum creatinine OR calculated* serum creatinine clearance (GFR can be used in place of creatinine or creatinine clearance) ≤ 1.5x upper limit of normal (ULN) OR ≥ 30 mL/min for participants with creatinine levels > 1.5x institutional ULN

         * Calculate serum creatinine clearance using the standard Cockcroft-Gault formula.

         Urine protein Urine dipstick for proteinuria < 2+ within 7 days prior to start of study treatment *Participants with ≥ 2+ proteinuria on dipstick analysis at baseline should undergo a 24-hour urine collection which must demonstrate < 1g of protein in 24 hours
      3. Hepatic - Serum total bilirubin ≤ 3 mg/dL , AST (SGOT) and ALT (SGPT) ≤ 5x ULN , Alkaline phosphatase (ALP) ≤ 8x ULN Coagulation - International Normalized Ratio (INR) or prothrombin time (PT) or activated partial thromboplastin time (aPTT) ≤ 2.0x ULN *This applies only to participants not receiving therapeutic anticoagulation; participants receiving therapeutic anticoagulation should be on a stable dose.

         Exclusion Criteria:

  <!-- -->

  1. Prior radiotherapy to the region of the liver that would result in excessive doses to normal tissues due to overlap of radiation therapy fields
  2. Prior selective internal radiotherapy/hepatic arterial Yttrium therapy, at any time
  3. Severe, active co-morbidity as per investigator
  4. More than five discrete intrahepatic parenchymal foci of definite HCC or left/right or main portal vein thrombus
  5. Direct tumor extension into the stomach, duodenum, small bowel or large bowel
  6. Measurable common or main branch biliary duct involvement with HCC
  7. Extrahepatic metastases or malignant nodes (that enhance with typical features of HCC) > 3.0 cm, in sum of maximal diameters (e.g. presence of one 3.4 cm metastatic lymph node or two 2 cm lung lesions).

     Note: benign non-enhancing periportal lymphadenopathy is not unusual in the presence of hepatitis and is permitted, even if the sum of enlarged nodes is > 2.0 cm.
  8. Prior liver transplant
  9. HIV positive
  10. Immunodeficiency requiring chronic systemic therapy or that may relapse
  11. Participants who have received prior immunotherapy.
  12. Participants with clinically meaningful ascites, defined as ascites requiring non-pharmacologic intervention (e.g. paracentesis) to maintain symptomatic control

      a. Note: Participants with ascites who require pharmacologic intervention (e.g. diuretics) to maintain symptomatic control and who have been on stable doses of diuretics for two months days prior to the first dose of study treatment are eligible.
  13. Participants with clinically meaningful encephalopathy
  14. Participants who have undergone prior solid organ or bone marrow transplant except for patients with prior renal transplant for whom dialysis may be employed in the event of graft rejection.
  15. Patients must have documented hepatitis virology status.

      a. Participants with active hepatitis B virus (HBV) infection must have a viral load < 500 IU/mL within 28 days prior to start of Tislelizumab and be on suppressive therapy (per local standard of care) for a minimum of fourteen days prior to start of study treatment and for the length of the study. b. Participants with co-infection with HBV and hepatitis C virus (HCV) are excluded.

      c. Participants with a history of HCV infection but with negative HCV RNA by PCR are considered non-infected with HCV and can enroll.
  16. Participants with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone are eligible.
  17. Participants with controlled Type 1 diabetes mellitus on a stable insulin regimen are eligible.
  18. Participants with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only are eligible provided: 1) rash covers < 10% of body surface area (BSA), disease is well controlled at baseline and requires only low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, flucinolone 0.01%, desonide 0.05%, aclometasone dipropionate 0.05%).
  19. Any malignancy ≤ 5 years before first dose of study drug except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated curatively (e.g. resected basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast).
  20. Treatment with a live, attenuated vaccine within four weeks prior to initiation of study treatment with Tislelizumab.

      1. Note: Seasonal vaccines for influenza and COVID-19 are generally inactivated vaccines and are allowed. Intranasal vaccines are live vaccines and are not allowed.
  21. Any condition that required systemic treatment with either corticosteroids (> 10 mg daily of prednisone or equivalent) or other immunosuppressive medication ≤ 14 days before first dose of study drug a. Note: Participants who are currently or have previously been on any of the following steroid regimens are not excluded: i. Adrenal replacement steroid (dose ≤ 10 mg daily of prednisone or equivalent) ii. Topical, ocular, intra-articular, intranasal, or inhaled corticosteroid with minimal systemic absorption iii. Short course (≤ 7 days) of corticosteroid prescribed prophylactically (e.g., for contrast dye allergy) or for the treatment of a non- autoimmune condition (e.g., delayed-type hypersensitivity reaction caused by contact allergen)
  22. With uncontrolled diabetes or > Grade 1 laboratory test abnormalities in potassium, sodium, or corrected calcium despite standard medical management or ≥ Grade 3 hypoalbuminemia ≤ 14 days before first dose of study drug
  23. With history of interstitial lung disease, non-infectious pneumonitis or uncontrolled diseases including pulmonary fibrosis, acute lung diseases, etc.
  24. With severe chronic or active infections requiring systemic antibacterial, antifungal or antiviral therapy, including tuberculosis infection, etc.
  25. Severe infections within 4 weeks before first dose of study drug, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia.
  26. Received therapeutic oral or intravenous antibiotics within two weeks before first dose of study drug
  27. Any major surgical procedure requiring general anesthesia ≤ 28 days before first dose of study drug
  28. Any of the following cardiovascular risk factors:

      a. Cardiac chest pain, defined as moderate pain that limits instrumental activities of daily living, ≤ 28 days before first dose of study drug b. Pulmonary embolism ≤ 28 days before first dose of study drug c. Any history of acute myocardial infarction ≤ 6 months before first dose of study drug d. Any history of heart failure meeting New York Heart Association (NYHA) Classification III or IV (Appendix 4) ≤ 6 months before first dose of study drug e .Any event of ventricular arrhythmia ≥ Grade 2 in severity ≤ 6 months before first dose of study drug f. Any history of cerebrovascular accident ≤ 6 months before first dose of study drug
  29. Has received any herbal medicine used to control cancer within fourteen days of the first study drug administration
  30. Participants with toxicities (because of prior anticancer therapy) which have not recovered to baseline or stabilized, except for AEs not considered a likely safety risk (e.g., alopecia, neuropathy and specific laboratory abnormalities)
  31. Underlying medical conditions (including laboratory abnormalities) or alcohol or drug abuse or dependence that, will be unfavorable for the administration of study drug or affect the explanation of drug toxicity or AEs or result in insufficient or might impair compliance with study c conduct.
  32. Concurrent participation in another therapeutic clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Safety as assessed by number of participants experiencing adverse events | 48 months
  Number of participants experiencing adverse events grade three or higher, as defined by Common Terminology Criteria for Adverse Events version 5.0 (NCI-CTCAE v5.0). Severity is a measure of intensity (eg, grade of a specific AE, mild [Grade 1], moderate [Grade 2], severe [Grade 3], or life-threatening [Grade 4]), whereas seriousness is classified by the criteria based on the regulatory definitions. Seriousness serves as the guide for defining regulatory reporting obligations from the Investigator Sponsor to applicable regulatory authorities as described in CTCAE version 5.0.

SECONDARY OUTCOMES:
Response and progression will be evaluated in this trial using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee (v1.1). | 48 months
  Changes in only the largest diameter (uni dimensional measurement) of the tumor lesions are used in the RECIST criteria.
  Measurable Disease:
  Tumor lesions: Must be accurately measured in at least 1 dimension (longest diameter in the plane of measurement is to be recorded) with a minimum size of:
  * 10 mm by CT scan (irrespective of scanner type) and MRI (no less than double the slice thickness and a minimum of 10 mm)
  * 10 mm caliper measurement by clinical exam (when superficial)
  * 20 mm by chest X ray (if clearly defined and surrounded by aerated lung) Malignant lymph nodes: To be considered pathologically enlarged and measurable, a lymph node must be ≥ 15 mm in short axis when assessed by CT scan (CT scan slice thickness recommended to be no greater than 5 mm). At baseline and in follow up, only the short axis will be measured and followed.

CONTACTS AND LOCATIONS:
Overall Officials: Salma Jabbour, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (2):
- United States (2):
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Montefiore Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No